CLINICAL TRIAL: NCT02007837
Title: Prospects for the Prevention of Pregnancy-induced Hypertension and Preeclampsia (4P) - a Randomised, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Prospects for the Prevention of Pregnancy-induced Hypertension and Preeclampsia Trial
Acronym: 4P
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Ghana Health Services (Other Government); University of Ghana (Other)
Responsible Party: Principal Investigator, Joyce L. Browne, MD, MSc,PhD candidate, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GHS-ERC: 05/05/2012
Record Dates: First submitted 2013-11-26; First posted 2013-12-11 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Pregnancy Induced Hypertension
Keywords: pregnancy induced hypertension; gestational hypertension; pre-eclampsia; preeclampsia; hypertensive disorders in pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Combined aspirin and multinutrient supplement (Experimental): In a single capsule, the following will be combined: 80mg low-dose aspirin, 1.2 grams calcium, 600 IU vitamin D, 5mg folic acid and 1000 ug vitamin B12
  Interventions: Drug: Combined aspirin and multinutrient supplement; Other: Daily text reminder text messages
- Placebo (Placebo Comparator): 5mg folic acid, cellulose filler
  Interventions: Other: Daily text reminder text messages

INTERVENTIONS:
Drug: Combined aspirin and multinutrient supplement — Single capsule with 80mg low-dose aspirin, 1.2 grams calcium, 600 IU vitamin D, 5mg folic acid and 1000 ug vitamin B12 mixed.
  Arms: Combined aspirin and multinutrient supplement
Other: Daily text reminder text messages

SUMMARY:
Hypertensive disorders of pregnancy (HDP) are with 50.000 deaths every year one of the major causes of maternal mortality worldwide, especially in low and middle income countries. This trial aims to determine whether a daily dose of combined low-dose aspirin, calcium, vitamin D3, folic acid and vitamin B12 in pregnancy reduces the incidence of pregnancy-induced hypertension in women at risk. Secondary and tertiary objectives include other maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* <16 weeks of gestation and over 18 years of age,
* Intention to have subsequent antenatal visits and delivery at the same clinic.
* Can receive text messages by phone or through the phone of a proxy.
* A moderate to high risk (>20%) of developing PIH

Exclusion Criteria:

* Pre-existing hypertension or hypertension before 20 weeks gestation.
* Likely non-compliance with the protocol in view of the treating physician
* Comorbidity interfering with the protocol
* Known contraindications to Investigational Product components

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 440 (Estimated)
Dates: Start 2018-01; Primary Completion 2018-04 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Development of pregnancy-induced hypertension (PIH) in pregnancy | up to 2 days after delivery.
  Development of a de novo systolic blood pressure (SBP) of > 140 mmHg, diastolic blood pressure (DBP) of >90 mmHg, measured at least twice.

SECONDARY OUTCOMES:
Maternal/obstetric outcomes | 6-16 weeks gestation, 16-24 weeks gestation, 26-36 weeks gestation, delivery and first days after
  maternal death, preeclampsia, eclampsia, hemolysis, elevated liver enzymes, and low platelet count (HELLP) syndrome, hemorrhage, caesarian section, other complications during pregnancy or delivery
Neonatal and infant outcomes | 6-16 weeks gestation, 16-24 weeks gestation, 26-36 weeks gestation, delivery and first days after
  preterm birth, Intra uterine death, stillbirth, neonatal mortality, congenital abnormality, Neonatal Intensive Care Unit (NICU) admission or pediatrician referral, birth weight, small for gestational age, apgar scores, other adverse effects. Infant outcomes: weight and height, health, occurrence of disease and general health status
Number of participants with (severe) adverse events as a measure of safety and tolerability | 1 year
  Number of patients with (severe) adverse events. Adverse events include any undesirable experience associated with the use of a medical product. Related to the product, bleeding incidences (including bruises), nausea, vomiting, will be explicitly reported.
  Severe adverse events are: death, life-threatening conditions, (prolonged) hospitalization, disability and permanent damage to mother or fetus, congenital abnormality, or other important (serious) medical events.

CONTACTS AND LOCATIONS:
Overall Officials: Diederick E Grobbee, MD PhD, Principal Investigator — UMC Utrecht; Patrick Frimpong, MBbCh, Principal Investigator — Ghana Health Services; Emmanuel K Srofenyoh, MBbCb, Principal Investigator — Ghana Health Services
Locations (2):
- Ghana (2):
  - La General Hospital, Accra
  - Ridge Regional Hospital, Accra